CLINICAL TRIAL: NCT01610154
Title: Contribution of Pancreatic αcells Function to Blood Glucose Regulation in Chinese Type 2 Diabetics- the Effect of Sitagliptin on Glucagon Secretion, Insulin Secretion and Insulin Resistance in Chinese Type 2 Diabetics
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Guangwei Li (Other)
Responsible Party: Sponsor-Investigator, Guangwei Li, director of endocrinology and cardiovascular disease center of Fuwai hospital, Chinese Academy of Medical Sciences, Fuwai Hospital
Organization: Chinese Academy of Medical Sciences, Fuwai Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CIFuwaiHospital-MISP39889
Record Dates: First submitted 2012-05-30; First posted 2012-06-01 (Estimated); Results first posted 2017-04-04 (Actual); Last update posted 2017-05-11 (Actual); Status verified 2017-04

CONDITIONS: Insulin Secretion; Insulin Resistance
Keywords: glucagon; dipeptidyl peptidase-4 inhibitor
MeSH Terms: conditions — Insulin Resistance | interventions — Sitagliptin Phosphate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Sitagliptin treatment (Experimental)
  Interventions: Drug: Sitagliptin

INTERVENTIONS:
Drug: Sitagliptin — Sitagliptin 100 mg QD for 12 weeks

SUMMARY:
1. The purpose of this study is to determine whether Sitagliptin therapy suppress glucagon release and improve glucose control in Chinese type 2 diabetic.
2. There are different effects of Sitagliptin therapy on blood glucose regulation, pancreatic alpha & beta cell function are different in lean (BMI<25) and overweight (BMI>25) Chinese type 2 diabetics.
3. The purpose of this study is to determine whether glucagon release may contribute over 30% to the hyperglycemia in Chinese type 2 diabetics.

ELIGIBILITY:
Inclusion Criteria:

1. Age: 25~60 years
2. Duration of disease < 3 years,no drug treatment for diabetes
3. Newly diagnosed type 2 diabetic patients (fasting plasma glucose > 7.0mmol/L or/and 2h postprandial blood glucose>11.1mmol/L WHO 1999)
4. Fasting plasma glucose < 10 mmol/L

Exclusion Criteria:

1. Type 1 diabetes
2. DKA, infection and other stress status
3. Autoimmune disease
4. Hepatic and renal diseases

Ages: 25 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 85 (Actual)
Dates: Start 2012-10; Primary Completion 2014-08 (Actual); Study Completion 2015-06 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Fuwai Hospital, Beijing, China

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Sitagliptin 100 mg QD for 12 weeks and followed-up every 4 weeks
Groups:
- Sitagliptin Treatment: Sitagliptin 100 mg QD for 12 weeks
Period: Overall Study
Arm/Group | Sitagliptin Treatment
Started | 85
Completed | 84
Not Completed | 1

BASELINE CHARACTERISTICS:
Arm/Group | Sitagliptin Treatment
Number analyzed (Participants) | 84
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 84
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.8 (12.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 37
  Male | 47
Region of Enrollment [Number; unit: participants]
  China | 84
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m2] | 25.8 (3.41)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Hemoglobin A1c (HbA1c)
Time Frame: Baseline to 12 weeks
Measure: Mean (Standard Deviation); unit: percentage
Groups:
- Sitagliptin: Sitagliptin 100 mg QD
Arm/Group | Sitagliptin
Number analyzed (Participants) | 84
percentage | -1.08 (0.13)

2. Secondary Outcome: Change From Baseline in Fasting Plasma Glucose (FPG)
Time Frame: Baseline to 12 weeks
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Sitagliptin
Number analyzed (Participants) | 84
mmol/L | -1.99 (0.18)

3. Secondary Outcome: Change From Baseline in Postprandial Plasma Glucose (PPG)
Time Frame: Baseline to 12 weeks
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Sitagliptin
Number analyzed (Participants) | 84
mmol/L | -4.69 (0.41)

4. Secondary Outcome: Change From Baseline in Insulin Sensitivity
Description: The insulin sensitivity was detected by evaluating the glucose infusion rate (GIR) with euglycemic hyperinsulinemic clamp test.
Time Frame: Baseline to 12 weeks
Measure: Median (Inter-Quartile Range); unit: mg/kg/min
Arm/Group | Sitagliptin
Number analyzed (Participants) | 84
mg/kg/min | 0.64 [0.27 to 1.58]

5. Secondary Outcome: Change From Baseline in Insulin Sensitivity in Patients With Different BMI
Description: as for outcome 4
Time Frame: Baseline to 12 weeks
Measure: Median (Inter-Quartile Range); unit: mg/kg/min
Groups:
- Non-obese Group: BMI<25 kg/m2
- Obese Group: BMI≥25 kg/m2
Arm/Group | Non-obese Group | Obese Group
Number analyzed (Participants) | 34 | 50
mg/kg/min | 0.42 [0.14 to 1.25] | 0.72 [0.32 to 1.93]

6. Secondary Outcome: Change From Baseline in Pancreatic β Cell Function
Description: The early phase insulin response (△I30/△G30) was adopted to determine β cell function.
Time Frame: Baseline to 12 weeks
Measure: Median (Inter-Quartile Range); unit: μu/ml/mmol
Arm/Group | Sitagliptin
Number analyzed (Participants) | 84
μu/ml/mmol | 2.53 [0.78 to 5.64]

7. Secondary Outcome: Change From Baseline in Pancreatic β Cell Function in Patients With Different BMI
Description: The early phase insulin response (△I30/△G30) was adopted to determine β cell function.
Time Frame: Baseline to 12 weeks
Measure: Median (Inter-Quartile Range); unit: μu/ml/mmol
Arm/Group | Non-obese Group | Obese Group
Number analyzed (Participants) | 34 | 50
μu/ml/mmol | 2.30 [0.96 to 4.65] | 2.85 [0.81 to 6.47]

8. Secondary Outcome: Change From Baseline in Pancreatic α Cell Function
Description: The glucagon-AUC was adopted to show pancreatic α cell function.
Time Frame: Baseline to 12 weeks
Measure: Mean (Standard Deviation); unit: min∙pg/ml
Arm/Group | Sitagliptin
Number analyzed (Participants) | 84
min∙pg/ml | -27.8 (32.3)

9. Secondary Outcome: Change From Baseline in Pancreatic α Cell Function in Patients With Different BMI
Description: The glucagon-AUC was adopted to show pancreatic α cell function.
Time Frame: Baseline to 12 weeks
Measure: Mean (Standard Deviation); unit: min∙pg/ml
Arm/Group | Non-obese Group | Obese Group
Number analyzed (Participants) | 34 | 50
min∙pg/ml | 13.6 (87.4) | -54.0 (307.4)

ADVERSE EVENTS:
Groups:
- Sitagliptin Treatment: Sitagliptin 100 mg QD
Arm/Group | Sitagliptin Treatment
Serious Adverse Events (participants affected / at risk) | 0/84
Other Adverse Events (participants affected / at risk) | 8/84
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sitagliptin Treatment (N=84)
Hypoglycemia ( symptom only) (Metabolism and nutrition disorders) | 5 (5)
Upper respiratory infection (Infections and infestations) | 1 (1)
Nasopharyngitis (Infections and infestations) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes